CLINICAL TRIAL: NCT04570059
Title: Effect of Information Promoting Textured Food Introduction on Parental Practices and Children Acceptance of Textured Foods
Brief Title: Textured Food Introduction Information and Parental Feeding Practices
Acronym: PATATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: UMR SayFood, Massy, France (Unknown); Funding from Carnot Qualiment (Project PATATE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ID RCB 2016-A00839-42
Record Dates: First submitted 2020-09-15; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Feeding Practices; Food Acceptance
Keywords: children; parental feeding practices; food texture; food oral processing; complementary feeding; recommendation

STUDY DESIGN:
Intervention Model Description: Intervention run between 8 and 15 months of the children, randomisation of children within a control (n=30) or intervention group (n=30).
Who Masked: Participant, Investigator
Masking Description: Parents are informed that the aim of the study was about the effect of complementary feeding recommendations on their child's eating behaviour but they are unaware of the focus on texture. They are also blinded to the group (intervention vs. control) to which they were allocated. This information is revealed to them after the end of the study. The principal investigator analyse the data without information on children allocation and groups effect are initially assessed without identification of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention program (Experimental): Intervention group
  Interventions: Behavioral: Counselling on textured food introduction between 8 and 15 months
- Usual Care (Active Comparator): Control group
  Interventions: Behavioral: Counselling on textured food introduction between 8 and 15 months

INTERVENTIONS:
Behavioral: Counselling on textured food introduction between 8 and 15 months — Intervention program : Advice and tips on the why and how introducing textured food during complementary feeding are grouped in a booklet and provided to participants. Monthly counselling via phone call by a dietician (at 9, 10, 11,12, 13, 14 months) and two baskets containing food preparation utensils and commercial textured foods provided at 8 and 12 months.
  Usual care : reflects the standard information provided within French national guidelines (PNNS). Two phone calls at 9 and 13 months. If questions are raised by parents, dieticians will restrict their responses based on the food guides of the PNNS. Two gift boxes containing presents for the child of same financial value as those provided to intervention group, provided at 8 and 12 months.
  Other Names: Food provision

SUMMARY:
The purpose of this study is to conduct an intervention with 60 parents of 8 months old children to test the effect of recommendations, compared to usual care, promoting the introduction of textured foods between 8 and 15 months on parental practices of use of textured foods and the effect of such practices on children acceptance for a variety of textured foods.

DETAILED DESCRIPTION:
The intervention tests the effect of providing parents with recommendations on textured food introduction between 8 and 15 months on their practices of offering of textured foods and their child's acceptance of textured foods. The intervention consists of advice and tips on the why and how introducing textured food during complementary feeding, which were not address in French national guidelines (Programme National Nutrition Santé (PNNS)) at the start of the study. Advise were developped from current literature knowledge and recommendations in other countries. They are accompanied with monthly counselling via phone calls by dietician and two baskets containing food preparation utensils and commercial textured foods. The intervention group (n=30) benefits from this intervention. The control group (n=30) receive general information on healthy eating provided by the food guides of the PNNS, phone calls collecting general information and 2 baskets containing baby gifts.

Acceptance is evaluated experimentally pre and post intervention in a laboratory setting evaluating children swallowing foods of different textures.

ELIGIBILITY:
Inclusion Criteria:

* parents ages ≥ 18 years old
* children born full term (≥37 weeks) and with weight ≥2500 g
* children introduced to complementary feeding after 4 months and before 6 months

Exclusion Criteria:

* children with episode of tube feedings, chronic disease, allergy and gastroesophageal reflux requiring medication
* children introduced to complementary feeding with baby-led weaning method
* children already involved in another study on eating behaviour

Ages: 1 Month to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Food texture exposure score | End of intervention (15 months)
  Food texture introduction assessed using a questionnaire developed to characterize the pattern of food texture exposure in French children aged 4-36 months (Demonteil et al., 2018). This questionnaire is composed of 188 items representing 61 foods commonly used in France in different texture combinations (puree, pieces, raw, cooked, etc.). Each food-texture combination present in the questionnaire is classified into one of three texture levels: 'purees' (soft and rough; T1 texture level), 'small/soft pieces' (T2 texture level) and 'hard/big pieces and double texture' (T3 texture level) . The number of introduced items is evaluated for each texture level (T1, T2 and T3), and a global child exposure score (TexExp) is calculated from the sum of all introduced items.
Textured food acceptance: scale | Pre and post intervention (8 and 15 months)
  Food texture acceptance is assessed during lab experiments. At each age, children participate in two experimental sessions in which they are offered several foods varying in texture. For each age, for a given child, the two sessions are planned during the same week. During one session, four different foods are offered to the child. Three trials of each food is run, trial offering is stopped after three consecutive refusals is emitted by the child. Experimenter evaluate whether the child swallow the trial. Acceptance is determined for each food as % of trial swallowed. Global acceptance outcome is calculated as the sum of frequency observed for each food.
  Parents evaluate the infant's liking of the food on a linear scale for each food trial.
  At the end of intervention, acceptance for 2 commercial baby food products is assessed by parents in home-setting. The parent records the weight of food eaten (g) and children 's liking of this food on a 9 point scale.

SECONDARY OUTCOMES:
Other maternal feeding practices | end of intervention (15 months)
  At the end of intervention, parents report if they search for information on texture introduction during the study. The type of foods offered (home-made or commercial foods), sharing meal with family and their motivation when buying food is assessed using dedicated questionnaires.
  A post-intervention interviews, organized after the end of the study allow to debrief with participants on their study participation.
Child feeding skills | Pre and post intervention (8 and 15 months)
  During the experimental session aiming at evaluating acceptance, the experimenter evaluate a set of behaviours : 'looks at the food', 'manipulate the food with fingers', 'puts the foods in the mouth with fingers/spoon', 'sucking', 'gagging', 'chewing', 'coughing/risk of chocking', 'has difficulties wih the food'.
  Parents will report children general feeding skills (holding a spoon in the mouth alone, eating with fingers, self-feeding with a fork, gagging) on a 4-point scale.
Number of teeth | Pre and post intervention (8 and 15 months)
  Parents report the number of teeth visible in their child mouth
Children chewing efficiency | Pre and post intervention (8 and 15 months)
  Determined during experimental session from children's ability to comminute a model gel. The gel is inserted in a mesh feeder and offered to the child for a 60s oral processing duration. Gel particles are collected from the feeder and photographed. The number of formed particles is used as marker of chewing efficiency.
Salivary flow rate | Pre and post intervention (8 and 15 months)
  Measured during experimental session using a cotton swab method (Salivette®, Sarsedt) for a 45-sec duration. Saliva collection was realized by the parent maintaining the swab for 45 seconds in child's mouth. The weight of the swab (g) is determined before and after collection and the exact exposure time (sec) is measured by the experimenter.
  Mesured weight and time are combined to determine flow rate (in g.min-1).
Children eating behaviour | 12 months
  Parent-reports using a Child Eating Behaviour Questionnaire adapted for toddlers (CEBQ-T) which is a validated questionnaire. The questionnaire is composed of 31 items. Parent answers to each item using a 6 category scale (never, rarely, sometimes, often, always, I don't know).The items are then grouped to define 7 dimensions : 'food responsiveness', 'enjoyment of food', 'satiety responsiveness', 'food fussiness', 'slowness in eating', 'emotional over-eating', and 'external food cue responsiveness'.Higher scores mean higher behaviours.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Tournier, PhD, Principal Investigator — INRAE UMR CSGA
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demonteil L, Ksiazek E, Marduel A, Dusoulier M, Weenen H, Tournier C, Nicklaus S. Patterns and predictors of food texture introduction in French children aged 4-36 months. Br J Nutr. 2018 Nov;120(9):1065-1077. doi: 10.1017/S0007114518002386. Epub 2018 Sep 11. PMID 30203737
- [Background] Tournier C, Demonteil L, Canon F, Marduel A, Feron G, Nicklaus S. A new masticatory performance assessment method for infants: A feasibility study. J Texture Stud. 2019 Jun;50(3):237-247. doi: 10.1111/jtxs.12388. Epub 2019 Feb 3. PMID 30667063
- [Background] Demonteil, L., et al. (2019).Longitudinal study on acceptance of food textures between 6 and 18 months. Food Quality and Preference 71: 54-65.
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- Available data/document: intervention material: Booklet of recommendation — https://hal.archives-ouvertes.fr/ — Booklet of recommendation provided to the intervention group (in French)